CLINICAL TRIAL: NCT00278629
Title: Non-myeloablative Autologous Hematopoietic Stem Cell Transplantation in Patients With Chronic Inflammatory Demyelinating Polyneuropathy: A Phase II Trial
Brief Title: Hematopoietic Stem Cell Transplantation in Chronic Inflammatory Demyelinating Polyneuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU FDA CIDP.AUTO2003
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-06

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hematopoietic Stem Cell Transplantation in CIDP (Experimental): Autologous hematopoietic stem cell transplantation will be performed after conditioning regimen of cyclophosphamide 200 mg/kg/intravenously(IV), rATG(thymoglobulin) 5.5 mg/kg/IV and rituximab 1000mg/IV.
  Interventions: Biological: hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: hematopoietic stem cell transplantation — Autologous hematopoietic stem cell transplantation

SUMMARY:
Chronic inflammatory demyelinating polyneuropathy is disease believed to be due to immune cells, cells which normally protect the body, but are now attacking the nerves in the body. As a result, the affected nerves fail to respond, or respond only weakly, to stimuli causing numbing, tingling, pain, and progressive muscle weakness.The likelihood of progression of the disease is high. This study is designed to examine whether treating patients with high dose cyclophosphamide (a drug which reduces the function of the immune system) and ATG (a protein that kills the immune cells that are thought to be causing disease), followed by return of the previously collected blood stem cells will stop the progression of CIDP. Stem cells are undeveloped cells that have the capacity to grow into mature blood cells, which normally circulate in the blood stream. The purpose of the high dose cyclophosphamide and ATG is to destroy the cells in the immune system. The purpose of the stem cell infusion is to evaluate whether this treatment will produce a normal immune system that will no longer attack the body.

DETAILED DESCRIPTION:
Selection of the Regimen for Immunosuppressive Therapy

Cyclophosphamide with ATG is a common conditioning regimen with two decades of experience in the treatment of aplastic anemia, and has been used safely without reported mortality in the treatment of autoimmune diseases such as systemic lupus erythematosus and rheumatoid arthritis.Cy / ATG is not associated with late malignancies or cataracts. Both cyclophosphamide and anti-thymocyte globulin (horse or rabbit ATG) are potent immunosuppressive agents. ATG contributes additional immunosuppression without additional cytotoxicity. ATG given shortly pre-transplant will contribute to the elimination of host T lymphocytes that survive cyclophosphamide SLE, an autoimmune disease responsive to cyclophosphamide, responds well to a CY / ATG conditioning regimen, but we have recently found that patients with either systemic lupus erythematosus (SLE) or neuromyelitis optica respond faster and may have more durable remissions to a regimen of "rituxan sandwich" in which rituxan is infused before and after standard cytoxan, rATG. For these reasons, "rituxan sandwich" will be the conditioning regimen utilized in this study.

5.2 Method of Harvesting Stem Cells

Based on the experience of the pilot studies, the current protocol will mobilize stem cells with granulocyte-colony stimulating factor (G-CSF) and collect stem cells by apheresis, with subsequent bone marrow harvest performed only if needed to supplement the peripheral blood stem cells (PBSC). Based on experience of autoimmune flares in patients receiving G-CSF alone for mobilization, patients will be mobilized with cyclophosphamide 2.0 g/m2 and G-CSF 5-10 mcg/kg.

5.3 Cyclophosphamide

Cyclophosphamide (CY) is an active agent in patients with a wide variety of malignancies. It is used frequently in the therapy of lymphoid malignancies and has potent immunosuppressive activity. It is frequently used as a cytotoxic and immunosuppressive agent in patients undergoing marrow transplants and as a treatment for patients with autoimmune diseases. It is an alkylating agent that requires hepatic metabolism to the active metabolites, phosphoramide mustard and acrolein. These active metabolites react with nucleophilic groups. It is available as an oral or intravenous preparation. Bioavailability is 90% when given orally. The half-life of the parent compound is 5.3 hours in adults, and the half-life of the major metabolite phosphoramide mustard is 8.5 hours. Liver or renal dysfunction will lead to prolonged serum half-life. CY is administered intravenously at a dosage of 50 mg/kg on each of 4 successive days (use adjusted ideal body weight if patient's actual body weight is greater than 100% ideal body weight). The major dose limiting side effect at high doses is cardiac necrosis. Hemorrhagic cystitis can occur and is mediated by the acrolein metabolite.This can be prevented by co-administration of MESNA or bladder irrigation. Other notable side effects include nausea, vomiting, alopecia, myelosuppression and SIADH. Refer to institutional manuals for more information about administration, toxicity and complications.

5.4 Rabbit-Derived Anti-Thymocyte Globulin (rATG)

Rabbit-derived anti-human thymocyte globulin (rATG) is a gamma globulin preparation obtained from hyperimmune serum of rabbits immunized with human thymocytes. rATG has been used predominately in solid organ transplant immunosuppressive regimens. rATG is a predominantly lymphocyte-specific immunosuppressive agent. It contains antibodies specific to the antigens commonly found on the surface of T cells. After binding to these surface molecules, rATG promotes the depletion of T cells from the circulation through mechanisms which include opsonization and complement-assisted, antibody-dependent, cell-mediated cytotoxicity. The plasma half-life ranges from 1.5 12 days. rATG is administered intravenously at a dose of 0.5 mg/kg recipient body weight on day -6 and at a dose of 1.0 mg/kg recipient body weight on days -5, -4, -3, -2, and -1. Unlike equine ATG, rabbit ATG does not require a pre-infusion skin test to check for hypersensitivity. Methylprednisolone 250 mg will be given before every dose of rATG. Additional medications such as diphenhydramine may be given at the discretion of the attending physician. Although rare, the major toxicity is anaphylaxis; chills, fever, pruritus or serum sickness may occur.

5.5 Rituxan Rituximab is a chimeric monoclonal antibody used in the treatment of B cell non-Hodgkin's lymphoma, B cell leukemia, and numerous autoimmune disorders. The recommended adult dosage for patients with low grade or follicular non-Hodgkin's lymphoma (NHL) is 375 mg/m2 infused intravenously and for adult patients with autoimmune diseases a standard 500 mg is generally given intravenously. The infusion may be given at weekly intervals for four total dosages or once every 2 weeks and repeated 2-3 times. Acetaminophen and diphenhydramine hydrochoride are given 30-60 minutes before the infusion to help reduce side effects. If given as a retreatment the dosage is the same. The majority of side effects occur after or during the first infusion of the drug. Some common side effects include dizziness, feeling of swelling of tongue or throat, fever and chills, flushing of face, headache, itching, nausea and vomiting, runny nose, shortness of breath, skin rash, and fatigue.

ELIGIBILITY:
Inclusion criteria:

* Definite CIDP according to the European Federation of Neurological Societies/Peripheral Nerve Society (EFNS/PNS) criteria

AND

* Clinically typical or atypical CIDP

AND

* Failure to tolerate or respond to, or an incomplete response to, or relapse after at least 3 months of conventional treatment consisting of corticosteroids (equivalent dosage of prednisone 1.0/mg/day to 0.75mg/kg/day to start with adequate tapering trials of no less than 0.5mg/kg/day), and/or either intravenous immunoglobulin (IVIg) or plasmapheresis or cytoxan or rituxan
* Failure to respond to therapy is defined by:

  1. Persistent muscle weakness Grade 3/5 or worse (MRC) in at least one muscle or grade 4/5 in at least two muscle groups OR
  2. Persistent dysphagia documented by either aspiration or insufficient clearing on videofluoroscopic examination.

     OR
  3. Persistent incapacitating sensory loss (e.g. gait ataxia, falls > 1/month)

     AND
  4. If patients are on IVIG or plasmapheresis, neurologic condition is documented to deteriorate (for example, new or increase finger tip paresthesias or increased leg heaviness) upon stopping IVIG (or plasmapheresis)@
* Monoclonal gammopathy of undetermined significance (MUGS) (in which the pathogenesis of are thought to be the same as CIDP) will be allowed provided bone marrow aspirate and biopsy rules out multiple myeloma.
* Other immune mediated or suspected immune mediated neuropathies such as multifocal motor neuropathy or anti-myelin-associated glycoprotein (anti-MAG) neuropathy may be treated but will be analyzed and reported separately.

Exclusion Criteria:

* Any evidence of hereditary cause for neuropathy that is known or likely hereditary demyelination neuropathy because of family history, foot deformity, mutilation of hands or feet, retinitis pigmentosa, ichthyosis, or liability to pressure palsies.
* Diphtheria, drug, or toxin exposure likely to be cause of neuropathy
* Conditions in which the pathogenesis of the neuropathy may be different from CIDP such as: Lyme disease (Borrelia burgdorferi infection), POEMS syndrome, Osteosclerotic myeloma, malignancies such as Waldenstrom macroglobulinemia, and Castleman's)
* Multiple myeloma
* HIV positive
* Insulin dependent Diabetes mellitus
* Chronic active hepatitis
* Age > 65 years old or < 18 years old
* Significant end organ damage such as (not caused by CIDP):

  1. Left ventricular ejection fraction (LVEF) <40% or deterioration of LVEF during exercise test on multigated acquisition scan (MUGA) or echocardiogram.
  2. Untreated life-threatening arrhythmia.
  3. Active ischemic heart disease or heart failure or myocardial infarction within the last 6 months
  4. Diffusing capacity of lung for carbon monoxide (DLCO) <40% or forced expiratory volume at one second (FEV1) / forced expiratory volume (FEV) < 50%
  5. Serum creatinine >2.0.
  6. Liver cirrhosis, transaminases > 2 x of normal limits or bilirubin >2.0 unless due to Gilbert disease.
* Prior history of malignancy except localized basal cell or squamous skin cancer or other localized cancer considered cured only by surgery
* Positive pregnancy test, inability or unwillingness to pursue effective means of birth control, or failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
* Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
* Inability to give informed consent.
* Major hematological abnormalities such as platelet count less than 100,000/ul or absolute neutrophil count (ANC) less than 1000/ul.
* Failure to collect at least 2.0 x 106 cluster of differentiation 34 (CD34+) cells by apheresis and, if necessary, bone marrow harvest is a contraindication to treatment, i.e., receiving the conditioning regimen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-02-21 (Actual); Primary Completion 2017-01-14 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Burt RK, Balabanov R, Tavee J, Han X, Sufit R, Ajroud-Driss S, Jovanovic B, Quigley K, Arnautovic I, Helenowski I, Sharrack B. Hematopoietic stem cell transplantation for chronic inflammatory demyelinating polyradiculoneuropathy. J Neurol. 2020 Nov;267(11):3378-3391. doi: 10.1007/s00415-020-10010-6. Epub 2020 Jun 27. PMID 32594300
- See also: Hematopoietic Stem Cell Transplantation for Chronic Inflammatory Demyelinating Polyradiculoneuropathy — https://doi.org/10.1007/s00415-020-10010-6

RESULTS

PARTICIPANT FLOW:
Groups:
- Hematopoietic Stem Cell Transplantation: Autologous hematopoietic stem cell transplantation will be performed after conditioning regimen of cyclophosphamide 200 mg/kg/intravenously(IV), rATG(thymoglobulin) 5.5 mg/kg/IV and rituximab 1000mg/IV.
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplantation
Started | 80
Completed | 66
Not Completed | 14
Not completed — Non-CIDP Immune-Mediated Peripheral Neur | 14

BASELINE CHARACTERISTICS:
Groups:
- Hematopoietic Stem Cell Transplantation for CIDP: Autologous hematopoietic stem cell transplantation will be performed after conditioning regimen of cyclophosphamide 200 mg/kg/intravenously(IV), rATG(thymoglobulin) 5.5 mg/kg/IV and rituximab 1000mg/IV.
Arm/Group | Hematopoietic Stem Cell Transplantation for CIDP
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants] — Population: The number analyzed differs from the overall because patients did not follow up and were subsequently excluded from the analysis.
  Participants
    number analyzed (Participants) | 60
    <=18 years | 0
    Between 18 and 65 years | 60
    >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] — Population: The number analyzed differs from the overall because patients did not follow up and were subsequently excluded from the analysis.
  years
    number analyzed (Participants) | 60
    (all) | 43 [20 to 63]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed differs from the overall because patients did not follow up and were subsequently excluded from the analysis.
  Participants
    number analyzed (Participants) | 60
    Female | 37
    Male | 23
Region of Enrollment [Number; unit: participants] — Population: The number analyzed differs from the overall because patients did not follow up and were subsequently excluded from the analysis.
  participants
    United States: number analyzed (Participants) | 60
    United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Survival
Description: Survival of participants who survived the treatment and up to 5 years post treatment.
Time Frame: up to 5 years
Population: The reason that the number analyzed is different from the overall number of participants anaylyzed is because 2 patients died from non treatment related conditions that were present before the transplant. Both deaths occurred more than 100 days after the hospital discharge from treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplantation for CIDP
Number analyzed (Participants) | 66
Participants
  Treatment Survival | 66
  Post Treament Survival | 64

2. Secondary Outcome: Disease Improvement - Medication Free Remission
Description: Post transplant immune medication-free remission with stable or improving neurological exam
Time Frame: 6 months, 1, 2, 3, 4 and 5 years post transplant
Population: The number analyzed in one or more rows differs from the over all number because not all patients returned for follow up.
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplantation for CIDP
Number analyzed (Participants) | 60
participants
  6 months post transplant | 48
  1 year post transplant | 48
  2 years after transplant | 47
  3 years post transplant: number analyzed (Participants) | 59
  3 years post transplant | 45
  4 years post transplant: number analyzed (Participants) | 50
  4 years post transplant | 39
  5 years post transplant: number analyzed (Participants) | 42
  5 years post transplant | 35

3. Secondary Outcome: Disease Improvement - Ambulatory Assistance
Description: Disease Improvement - Requires No Assistance to Ambulate
Time Frame: pre transplant, 6 months, 1, 2, 3, 4 and 5 years post transplant
Population: The number analyzed in one or more rows differs from the overall number analyzed because not all patients returned for followed up testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplantation for CIDP
Number analyzed (Participants) | 60
Participants
  pre transplant | 19
  6 months post transplant | 41
  1 year post transplant | 49
  2 years post transplant: number analyzed (Participants) | 59
  2 years post transplant | 48
  3 years post transplant: number analyzed (Participants) | 59
  3 years post transplant | 48
  4 years post transplant: number analyzed (Participants) | 50
  4 years post transplant | 43
  5 years post transplant: number analyzed (Participants) | 42
  5 years post transplant | 35

4. Secondary Outcome: Change in Disability and Strength Functional Scales
Description: Change in the Medical Research Council (MRC) Scale: range is 0 (quadriplegic) - 60 (normal).
Time Frame: Pre Transplant, 6 months, 1, 2, 3, 4 and 5 years post transplant
Population: The reason the number analyzed in one or more rows differs from the overall number analyzed is because not all patients returned for followed up testing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hematopoietic Stem Cell Transplantation for CIDP
Number analyzed (Participants) | 60
score on a scale
  Pre Transplant | 51.8 (6.3)
  6 Months Post Transplant: number analyzed (Participants) | 50
  6 Months Post Transplant | 54.8 (5.6)
  1 year post transplant: number analyzed (Participants) | 45
  1 year post transplant | 57 (4.18)
  2 years post transplant: number analyzed (Participants) | 44
  2 years post transplant | 57 (4.3)
  3 years post transplant: number analyzed (Participants) | 39
  3 years post transplant | 57 (3.9)
  4 years post transplant: number analyzed (Participants) | 33
  4 years post transplant | 57 (3.9)
  5 years post transplant: number analyzed (Participants) | 26
  5 years post transplant | 57 (4.3)

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Hematopoietic Stem Cell Transplantation for CIDP
All-Cause Mortality (participants affected / at risk) | 2/66
Serious Adverse Events (participants affected / at risk) | 2/66
Other Adverse Events (participants affected / at risk) | 29/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation for CIDP (N=66)
Total Parenteral Nutrition - due to vomiting (Gastrointestinal disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Transient Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Non Transplant Related Death (Cardiac disorders) | 1 (1)
Non Transplant Related Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Gastric Cancer
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation for CIDP (N=66)
Hypophosphatemia (Metabolism and nutrition disorders) | 29 (29)
Febrile Neutropenia (General disorders) | 26 (26)
Hypokalemia (Metabolism and nutrition disorders) | 19 (19)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Infections (Infections and infestations) | 8 (8)
Clostridium Difficile Diarrhea (Infections and infestations) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes